CLINICAL TRIAL: NCT06403241
Title: The Association Between Food Timing and Composition on Gastrointestinal Injury, Stress Hormone and Gastrointestinal Complains in Elite Rowers After 2000m Ergometer Test - an Observational Study.
Brief Title: The Association Between Food Timing and Composition on Gastrointestinal Injury, Stress Hormone and Gastrointestinal Complains.
Status: Completed | Type: Observational
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Other Study IDs: Rowerscometetive2023
Record Dates: First submitted 2024-04-26; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2023-06

CONDITIONS: Endothelial Dysfunction
Keywords: athlete's diet; endotoxemia; cortisol; gut injury; gut permeability; exercise
MeSH Terms: conditions — Endotoxemia; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 2000 meter ergometer test — Rowers performed 2000m ergometer test.A 2,000-m time trial is a standard test used to assess performance in rowers.

SUMMARY:
The study aimed to check the influence of timing and composition of diet on markers of gut injury, endotoxemia and stress.

DETAILED DESCRIPTION:
The research protocol includes detailed food intake analysis, including timing and composition, markers related to the neuroendocrine pathway cortisol, and observations of individually experienced symptoms. Moreover, the study also explores intestinal injury and endotoxemia parameters, such as I-FABP, CLDN-3, and LBP. As a first goal, this study investigates the timing and composition of food intake concerning changes in gut integrity, cortisol levels, and gastrointestinal symptoms. Investigators explored whether an athlete's nutritional intake influences any GI disturbance induced by high-intensity exercise. As a second goal, Investigators tried to connect symptoms and markers from both pathways with gastrointestinal complaints. Investigators hypothesised that cortisol levels would be more profound than other studied parameters in gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Membership in Polish Rowing Team,
* minimum five years of training,
* total training time minimum of 240 minutes,
* filling out a food diary,
* finishing 2000-meter ergometer test.

Exclusion Criteria:

* Probiotics within the last three months,
* prebiotics within the last three months
* antibiotic therapy within the last three months,
* dietary regime,
* gastrointestinal diseases,
* lactose intolerance

Ages: 18 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male rowers age 18 - 22 years.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
I-FABP (intestinal fatty acid binding protein)to measure epithelial wall injury | Blood samples was taken from the cubital vein at three-time points: before each stress test (after overnight fasting) up to one hour after getting up, 1 minute after the test, and 1-hour recovery period
  I-FABP concentration measured in blood [ng/ml] using commercially available enzyme-linked immunosorbent assays
Claudin to measure tight junction leakage | Blood samples was taken from the cubital vein at three-time points: before each stress test (after overnight fasting) up to one hour after getting up, 1 minute after the test, and 1-hour recovery period
  Zonulin concentration measured in blood [ng/ml] using commercially available enzyme-linked immunosorbent assays
LBP (lipopolysaccharide binding protein) to measure endotoxin | Blood samples was taken from the cubital vein at three-time points: before each stress test (after overnight fasting) up to one hour after getting up, 1 minute after the test, and 1-hour recovery period
  LBP concentration measured in blood [ug/ml] using commercially available enzyme-linked immunosorbent assays
Lactic acid to measure fatigue after the race | Blood samples was taken from the cubital vein at three-time points: before each stress test (after overnight fasting) up to one hour after getting up, 1 minute after the test
  Lactate concentration measured in capillary blood from earlobe [mmol/L] using a commercially available kit (Diaglobal, Berlin, Germany)
Corisol | Blood samples was taken from the cubital vein at three-time points: before each stress test (after overnight fasting) up to one hour after getting up, 1 minute after the test, and 1-hour recovery period
  Stress hormoneconcentration measured in blood [ng/ml] using commercially available enzyme-linked immunosorbent assays

SECONDARY OUTCOMES:
energy | whole day (24hours) before test, in the morning before the test
  energy [kcal ]of food intake measured by food diary
protein | whole day (24hours) before test, in the morning before the test
  protein [g ]of food intake measured by food diary
fat | whole day (24hours) before test, in the morning before the test
  fat [g ]of food intake measured by food diary
carbohydrate | whole day (24hours) before test, in the morning before the test
  carbohydrate [g ]of food intake measured by food diary
glucose | whole day (24hours) before test, in the morning before the test
  glucose [g ]of food intake measured by food diary
lactose | whole day(24hours) before test, in the morning before the test
  lactose [g ]of food intake measured by food diary
saccharose | whole day (24hours) before test, in the morning before the test
  saccharose [g ]of food intake measured by food diary
fructose | whole day (24hours) before test, in the morning before the test
  fructose [g ]of food intake measured by food diary
fiber | whole day (24hours) before test, in the morning before the test
  fiber [g ]of food intake measured by food diary
Body mass | in the morning before the test up to 1 hour after getting up
  Body mass [kg] measured by electronic scale to the nearest 0,05 kg (Tanita BC 418 MA Tanita Corporation, Tokyo, Japan).
Body fat | in the morning before the test up to 1 hour after getting up
  Body fat [%] measured by electronic scale (Tanita BC 418 MA Tanita Corporation, Tokyo, Japan).
Total body water | in the morning before the test up to 1 hour after getting up
  Body fat [%] measured by electronic scale (Tanita BC 418 MA Tanita Corporation, Tokyo, Japan).
Lean body mass | in the morning before the test up to 1 hour after getting up
  Lean body mass [kg] measured by electronic scale (Tanita BC 418 MA Tanita Corporation, Tokyo, Japan).
height | in the morning before the test up to 1 hour after getting up
  [cm] measured by high meter
self reported gastrointestinal scale | up to 1 hours after the test
  10 point scale

CONTACTS AND LOCATIONS:
Overall Officials: Anna Skarpańska-Stejnborn, professor, Study Director — Poznan University of Physical Education
Locations (1):
- Poznan University of Physical Education, Faculty of Sport Sciences in Gorzow, Gorzów Wielkopolski, Lubusz Voivodeship, Poland